CLINICAL TRIAL: NCT03457142
Title: Phase II Study of Targeting CD28 in Multiple Myeloma With Abatacept (CTLA4-Ig) to Overcome Resistance to Chemotherapy
Brief Title: Abatacept, Ixazomib Citrate, and Dexamethasone in Treating Patients With Multiple Myeloma Resistant to Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding ended
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 47217; NCI-2017-02430 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 47217 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2018-02-27; First posted 2018-03-07 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Abatacept; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (abatacept, ixazomib citrate, dexamethasone) (Experimental): Patients receive abatacept IV over 30 minutes on day 1 of course 1, then SC on days 2, 8, 15, and 22 of course 1, and then on days 1, 8, 15, and 22 of subsequent courses. Patients also receive ixazomib citrate PO QD on days 1, 8, and 15 and dexamethasone on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Abatacept; Drug: Dexamethasone; Drug: Ixazomib Citrate; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Abatacept — Given IV and SC
  Other Names: BMS-188667; CTL A4-Ig B7 Inhibitor; CTLA4-Ig; cytotoxic T lymphocyte-associated antigen-4; Orencia; RG2077
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; Ninlaro
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well abatacept, ixazomib citrate, and dexamethasone work in treating patients with multiple myeloma that is resistant to chemotherapy. Abatacept may block certain proteins that are present on multiple myeloma cells that have been shown to protect against chemotherapy. Drugs used in chemotherapy, such as ixazomib citrate and dexamethasone, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving abatacept, ixazomib citrate, and dexamethasone may work better at treating patients with multiple myeloma resistant to chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the therapeutic efficacy (as measured by response rate) of abatacept + ixazomib citrate (ixazomib) + dexamethasone in multiple myeloma patients who have relapsed (or who are primary refractory) following treatment with their first proteasome inhibitor-containing regimen (excluding ixazomib), compared to historical controls of ixazomib + dexamethasone.

SECONDARY OBJECTIVES:

I. To assess the toxicity profile of abatacept + ixazomib + dexamethasone in multiple myeloma patients who have relapsed (or who are primary refractory) following treatment with their first proteasome inhibitor-containing regimen, compared to historical controls of ixazomib + dexamethasone.

II. To assess progression-free and overall survival profile of abatacept + ixazomib + dexamethasone in multiple myeloma patients who have relapsed (or who are primary refractory) following treatment with their proteasome inhibitor-containing regimen, compared to historical controls of ixazomib + dexamethasone.

TERTIARY OBJECTIVES:

I. Assess whether myeloma expression of CD28, CD86, serum kynurenine and/or IL-6 are correlated with specific clinical outcomes.

OUTLINE:

Patients receive abatacept intravenously (IV) over 30 minutes on day 1 of course 1, then subcutaneously (SC) on days 2, 8, 15, and 22 of course 1, and then on days 1, 8, 15, and 22 of subsequent courses. Patients also receive ixazomib citrate orally (PO) once daily (QD) on days 1, 8, and 15 and dexamethasone on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma who have relapsed (or who are primary refractory) following treatment with a proteasome inhibitor-containing regimen (excluding ixazomib) and who have not been treated with a second proteasome inhibitor (ixazomib, bortezomib, carfilzomib or other proteasome inhibitor).
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2 at study entry
* Must be free of systemic infection:

  * Subjects with active infections (whether or not they require antibiotic therapy) may be eligible after complete resolution of the infection
  * Subjects on antibiotic therapy must be off antibiotics for at least 7 days before beginning treatment
* Absolute neutrophil count >= 750/mm^3
* Platelet count >= 25,000/mm^3
* Creatinine clearance >= 30 mL/min
* Total bilirubin =< 3 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN
* Patient's multiple myeloma cells are positive for CD28 or CD86 expression by flow cytometry or immunohistochemistry (in any proportion) CD28 or CD86 positivity can have been determined on previous bone marrow aspirates or biopsies
* Disease free of prior malignancies for > 2 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma ?in situ? of the cervix or breast
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Prior treatment with ixazomib
* Inability to take ixazomib or abatacept
* Life expectancy less than 4 months
* Patients with a known diagnosis of plasma cell leukemia
* Known active tuberculosis or fungal infection
* Known seropositive for or active viral infection with, human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or, which confounds the ability to interpret data from the study
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator?s opinion deems the participant an unsuitable candidate to receive study drug
* Received an investigational agent within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2024-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hillengass, MD, PhD, Principal Investigator — Roswell Park Cancer Institute
Locations (3):
- United States (3):
  - Roswell Park Cancer Institute, Buffalo, New York
  - St. Francis Hospital, East Hills, New York
  - Good Samaritan Hospital, West Islip, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Abatacept, Ixazomib Citrate, Dexamethasone)
Started | 15
Completed | 14
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Abatacept, Ixazomib Citrate, Dexamethasone)
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of Abatacept + Ixazomib Citrate + Dexamethasone in Multiple Myeloma Patients
Description: Will be compared to historical controls of ixazomib citrate + dexamethasone. Responses to treatment will be measured by serum immunoglobulins, serum free kappa and lambda light chains, serum protein electrophoresis/immunofixation electrophoresis, and 24-hour urine protein electrophoresis/immunofixation. International uniform response criteria will be used. The anti-myeloma activity will be evaluated on an exploratory basis and will be summarized using descriptive statistics or graphical methods. No formal comparison will be carried forth.
Time Frame: 1 cycle of 28 days
Population: 1 patient experienced death prior to disease response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Abatacept, Ixazomib Citrate, Dexamethasone)
Number analyzed (Participants) | 14
Participants
  Complete Response | 1
  Partial Response | 4
  Stable Disease | 8
  Progressive Disease | 1

2. Secondary Outcome: Incidence of Adverse Events Assessed Using National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: The adverse events and drug related toxicities will be summarized by grade using frequencies and relative frequencies. The rate of grade 3 or higher toxicities that are probably or definitely related to abatacept will be reported with 90% confidence intervals obtained using Jeffrey?s prior method.
Time Frame: Up to 30 days after last dose
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Abatacept, Ixazomib Citrate, Dexamethasone)
Number analyzed (Participants) | 15
Participants | 5
Statistical Analysis 1: Comparison: Treatment (Abatacept, Ixazomib Citrate, Dexamethasone); Test type: Other — No formal test, a confidence interval estimate for the grade 3+ treatment related AE rate; grade 3+ treatment related AE rate = 0.33, 90% CI 2-sided [0.17 to 0.54]

3. Secondary Outcome: Overall Survival
Description: Defined as the time from treatment initiation until death or last follow-up. Will be summarized using standard Kaplan-Meier methods; where estimates of median survival and survival rates will be obtained with 90% confidence intervals.
Time Frame: From the date of the first study treatment until initiation of a new therapy, death, or end of follow-up (up to 5 years); whichever occurs first.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Abatacept, Ixazomib Citrate, Dexamethasone)
Number analyzed (Participants) | 15
months | 33.6 [14.5 to NA] — Insufficient number of events observed to calculate the upper bound for the 90% confidence interval.

4. Secondary Outcome: Progression-free Survival
Description: Defined as the time from treatment initiation until disease progression, death, or last follow-up. Will be summarized using standard Kaplan-Meier methods; where estimates of median survival and survival rates will be obtained with 90% confidence intervals.
Time Frame: From the date of the first study treatment to the date of first observed disease progression or death due to any cause, assessed up to 5 years
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Abatacept, Ixazomib Citrate, Dexamethasone)
Number analyzed (Participants) | 15
months | 11.1 [5.7 to 15.9]

5. Other Pre Specified Outcome: CD28 and CD86 Expression Assessed by Flow Cytometry
Description: The expression/levels and response will be evaluated using logistic regression models.
Time Frame: Up to 5 years
Population: These measurements were not collected and are not available for reporting.
Arm/Group | Treatment (Abatacept, Ixazomib Citrate, Dexamethasone)
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Serum Kynurenine and IL-6 Levels
Description: The association between CD28, CD86, serum kynurenine and IL-6 expression/levels and response will be evaluated using logistic regression models.
Time Frame: Up to 5 years
Population: These measurements were not collected and are not available for reporting.
Arm/Group | Treatment (Abatacept, Ixazomib Citrate, Dexamethasone)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were captured from the start of treatment until up to 30 days after the end of treatment; which ranged from 1.4 to 16.6 months (median = 6.8 months). All-cause mortality is captured for up to 5 years post treatment initiation.
Arm/Group | Treatment (Abatacept, Ixazomib Citrate, Dexamethasone)
All-Cause Mortality (participants affected / at risk) | 1/15
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Abatacept, Ixazomib Citrate, Dexamethasone) (N=15)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Abatacept, Ixazomib Citrate, Dexamethasone) (N=15)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Blurred vision (Eye disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 8 (8)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 6 (6)
Generalized edema (General disorders) | 2 (2)
Injection site reaction (General disorders) | 1 (1)
Joint infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Platelet count decreased (Investigations) | 3 (3)
Weight gain (Investigations) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Agitation (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (6)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Hot flashes (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT03457142/Prot_SAP_000.pdf